CLINICAL TRIAL: NCT01762046
Title: Study to Understand the Genetics of the Acute Response to Metformin and Glipizide in Humans
Acronym: SUGAR-MGH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Joslin Diabetes Center (Other); Broad Institute of MIT and Harvard (Other)
Responsible Party: Principal Investigator, Jose C. Florez, MD, PhD, Assistant Physician in Endocrinology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007p000193
Record Dates: First submitted 2012-12-28; First posted 2013-01-07 (Estimated); Results first posted 2024-05-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Pharmacogenetics; Genetics; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glipizide; Metformin; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glipizide and Metformin (Other): On day 1, subjects will receive a single oral dose of glipizide 5 mg, and will have blood drawn at various time points for up to 240 minutes. During study days 2-7, the participants will fill out a dietary intake food record, including 3 weekdays and one weekend day. During days 6-8, the subject will receive a short-course metformin treatment of four 500-mg doses. On the morning of study day 8, 60 minutes after taking the fourth metformin dose, the subject will do a 75g Oral Glucose Tolerance Test. Blood draws will again be taken at time points for 120 minutes.
  Interventions: Drug: Glipizide; Drug: Metformin; Other: Oral Glucose Tolerance Test

INTERVENTIONS:
Drug: Glipizide
Drug: Metformin
Other: Oral Glucose Tolerance Test

SUMMARY:
The SUGAR-MGH investigators are studying the influence of inherited gene variants on the response to two commonly prescribed type 2 diabetes medications, metformin and glipizide. They hypothesize that variants in genes that are associated with type 2 diabetes or related traits may impact the effect of anti-diabetic medications. In addition, physiological responses to an insulin secretagogue or an insulin sensitizer may shed light on the mechanism of action of reported genetic associations.

DETAILED DESCRIPTION:
Several common genetic variants have been reliably associated with type 2 diabetes and related glycemic traits. Study investigators hypothesize that variants in genes that are reproducibly associated with type 2 diabetes or related glycemic traits may impact the effect of anti-diabetic medications. In particular, sulfonylureas may have differential effects on individuals depending on the allelic variant they carry at KCNJ11 E23K; conversely, because TCF7L2 is postulated to influence insulin secretion by regulating the action of glucagon-like peptide 1 (GLP-1), and sulfonylureas act at a different step in the insulin secretion pathway, the effect of sulfonylureas on insulin secretion could be independent of genetic variation at TCF7L2. In addition, physiological responses to an insulin secretagogue or an insulin sensitizer may shed light on the mechanism of action of reported genetic associations.

Despite the convincing associations of several genetic variants with type 2 diabetes and their involvement in physiological pathways involved in drug response, their impact on pharmacological interventions has not been systematically examined. The completion of the Human Genome Project and the high-density characterization of common human variation in four different ethnic groups highlight the promise of genomic medicine. The elucidation of the genetic architecture of complex phenotypes may help clinicians understand disease heterogeneity, uncover new pathophysiological mechanisms, open the opportunity for novel therapeutic interventions, provide predictive diagnostic and prognostic information, and allow for individually tailored therapy that takes into account both the probability of response and the incidence of drug-induced complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female > 18 years of age
* Investigators will target preferentially people at risk of diabetes or requiring diabetes meds
* The first tier of risk will be illustrated by one of the following variables (e.g. established type 2 diabetes on diet therapy alone, elevated random glucose in electronic medical record, PCOS, metabolic syndrome, obesity, history of gestational diabetes, etc.)
* The second tier of risk will be illustrated by other features that correlate with diabetes risk, such as a history of hypertension or dyslipidemia
* Otherwise healthy subjects may also be candidates for the study.
* Able and willing to give consent relevant to genetic investigation

Exclusion Criteria:

* Pregnant, nursing or at risk of becoming pregnant
* Currently taking any medications for the treatment of diabetes
* Currently on metformin for any other indication (e.g. PCOS)
* Onset of diabetes in a family member before age 25, with autosomal transmission of diabetes across three generations
* History of liver or kidney disease
* Known severe allergic reactions to sulfonamides
* History of porphyria
* Documented estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m2, based on the most recent serum creatinine measurement available in the electronic medical record, and calculated by the Modification of Diet in Renal Disease equation (49) available at http://www.nephron.com/cgi-bin/MDRD_GFR.cgi
* Currently taking medications known to affect glycemic parameters, such as glucocorticoids, growth hormone or fluoroquinolones
* Planned radiologic or angiographic study requiring contrast within one week of completion of this study
* Established coronary artery disease (CAD), defined as:
* History of myocardial infarction.
* History of revascularization (coronary artery bypass grafting, percutaneous coronary intervention (e.g. stenting or balloon angioplasty).
* Evidence of ischemia on cardiac stress test.
* Enrolled in any other interventional study at time of screening through completion of study protocol
* History of bariatric surgery
* History of seizures
* History of stroke/CVA

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1033 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Florez, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts

REFERENCES:
- [Derived] Chen L, Li JH, Kaur V, Muhammad A, Fernandez M, Hudson MS, Goldfine AB, Florez JC. The presence of two reduced function variants in CYP2C9 influences the acute response to glipizide. Diabet Med. 2020 Dec;37(12):2124-2130. doi: 10.1111/dme.14176. Epub 2019 Nov 25. PMID 31709648
- [Derived] Srinivasan S, Kaur V, Chamarthi B, Littleton KR, Chen L, Manning AK, Merino J, Thomas MK, Hudson M, Goldfine A, Florez JC. TCF7L2 Genetic Variation Augments Incretin Resistance and Influences Response to a Sulfonylurea and Metformin: The Study to Understand the Genetics of the Acute Response to Metformin and Glipizide in Humans (SUGAR-MGH). Diabetes Care. 2018 Mar;41(3):554-561. doi: 10.2337/dc17-1386. Epub 2018 Jan 11. PMID 29326107
- [Derived] Walford GA, Colomo N, Todd JN, Billings LK, Fernandez M, Chamarthi B, Warner AS, Davis J, Littleton KR, Hernandez AM, Fanelli RR, Lanier A, Barbato C, Ackerman RJ, Khan SQ, Bui R, Garber L, Stolerman ES, Moore AF, Huang C, Kaur V, Harden M, Taylor A, Chen L, Manning AK, Huang P, Wexler D, McCarthy RM, Lo J, Thomas MK, Grant RW, Goldfine A, Hudson MS, Florez JC. The study to understand the genetics of the acute response to metformin and glipizide in humans (SUGAR-MGH): design of a pharmacogenetic resource for type 2 diabetes. PLoS One. 2015 Mar 26;10(3):e0121553. doi: 10.1371/journal.pone.0121553. eCollection 2015. PMID 25812009

RESULTS

PARTICIPANT FLOW:
Groups:
- Glipizide and Metformin: On day 1, subjects will receive a single oral dose of glipizide 5 mg, and will have blood drawn at various time points for up to 240 minutes. During study days 2-7, the participants will fill out a dietary intake food record, including 3 weekdays and one weekend day. During days 6-8, the subject will receive a short-course metformin treatment of four 500-mg doses. On the morning of study day 8, 60 minutes after taking the fourth metformin dose, the subject will do a 75g Oral Glucose Tolerance Test. Blood draws will again be taken at time points for 120 minutes.
  Glipizide
  Metformin
  Oral Glucose Tolerance Test
Period: Overall Study
Arm/Group | Glipizide and Metformin
Started | 1033
Completed | 1033
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 1033
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1033 subjects were enrolled and completed the study but some disqualified for various reasons like not fasting for the fasting visit due to having chewed gum, or having had black coffee, and in the end we have 1000 subjects with viable phenotype and genotype data.
  years
    number analyzed (Participants) | 1000
    (all) | 47.2 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 557
  Male | 476
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 229
  White | 702
  More than one race | 21
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 1033
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 1033 subjects completed the study but 33 subjects were disqualified for various reasons (such as: having chewed gum before the fasting visits, had coffee before the fasting visit etc.), and in the end we have 1000 subjects with viable phenotype and genotype data.
  kg/m^2
    number analyzed (Participants) | 1000
    (all) | 30.14 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Glipizide Response as Measured by Area Over the Glucose Curve Between Time 0 and 240 Minutes According to Genotype
Description: Investigators will measure glucose levels at 0,30,60,90,120,180 and 240 minutes post 5mg Glipizide administration on Visit 1(Day1), and compare them by genotype at selected loci.
Time Frame: 0, 30, 60, 90, 120, 180 and 240 minutes post 5mg oral glipizide dose, Day 1 (visit 1)
Population: 1000 subjects were genotyped for SNP rs7903146 (in the TCF7L2 gene). We are showing Area over the curve for glucose that was measured between time 0 to 240 minutes. 10 subjects didn't pass the QC for genotype analysis.
Measure: Mean (Standard Deviation); unit: mg/dl x time(minutes)
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 990
mg/dl x time(minutes)
  Area over the Glucose curve for TCF7L2 CC genotype: number analyzed (Participants) | 500
  Area over the Glucose curve for TCF7L2 CC genotype | 4893.5 (2079.4)
  Area over the Glucose curve for TCF7L2 CT genotype: number analyzed (Participants) | 400
  Area over the Glucose curve for TCF7L2 CT genotype | 5032.6 (2161)
  Area over the Glucose curve for TCF7L2 TT Genotype: number analyzed (Participants) | 90
  Area over the Glucose curve for TCF7L2 TT Genotype | 6011 (3204.8)

2. Primary Outcome: Glipizide Response as Measured by Area Under the Insulin Curve Between Time 0 and 240 Minutes According to Genotype
Description: Investigators will measure insulin levels at 0,30,60,90,120,180 and 240 minutes post 5mg Glipizide administration on Visit 1(Day1), and compare them by genotype at selected loci.
Time Frame: 0,30,60,90,120,180 and 240 minutes on Day 1 (Visit 1)
Population: 1000 subjects were genotyped for SNP rs7903146 (in the TCF7L2 gene). We are showing Area under the curve for Insulin that was measured between time 0 to 240 minutes. 10 subjects didn't pass the QC for genotype analysis.
Measure: Mean (Standard Deviation); unit: mU/L x time (minutes)
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 990
mU/L x time (minutes)
  Area under the InsulinCurve for TCF7L2 CC genotype: number analyzed (Participants) | 500
  Area under the InsulinCurve for TCF7L2 CC genotype | 1141 (1910)
  Area under the InsulinCurve for TCF7L2 CT genotype: number analyzed (Participants) | 400
  Area under the InsulinCurve for TCF7L2 CT genotype | 1278 (1455)
  Area under the InsulinCurve for TCF7L2 TT genotype: number analyzed (Participants) | 90
  Area under the InsulinCurve for TCF7L2 TT genotype | 1400 (1447)

3. Primary Outcome: Metformin Response - Change in Fasting Glucose From Visit 1 to Visit 2
Description: Investigators will measure the change in glycemic measures between Visit 1 (Day 1) and Visit 2 (Day 8) as an index of Metformin response, and compare them by genotype at selected loci. HOMA-IR is calculated from fasting glucose and fasting insulin values at both visit 1 (day 1) and visit 2 (day 8). HOMA-IR was calculated using (fasting glucose*fasting insulin)/405) formula.
Time Frame: Day 1 (Visit 1) and Day 8 (Visit 2)
Population: We looked at fasting glucose at Visit 2 minus fasting glucose at visit 1 to see if there are differences by genotype at rs7903146 after Metformin treatment in the 1000 subjects in this study. 10 subjects didn't pass the QC for genotype analysis.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 990
mg/dl
  FastingGlucose V2-FastingGlucose V1 in CC Genotype: number analyzed (Participants) | 500
  FastingGlucose V2-FastingGlucose V1 in CC Genotype | -2.1 (8.1)
  FastingGlucose V2-FastingGlucose V1 in CT Genotype: number analyzed (Participants) | 400
  FastingGlucose V2-FastingGlucose V1 in CT Genotype | -2.2 (8.2)
  FastingGlucose V2-FastingGlucose V1 in TT Genotype: number analyzed (Participants) | 90
  FastingGlucose V2-FastingGlucose V1 in TT Genotype | -6.1 (11)

4. Primary Outcome: Metformin Response - Change in HOMA-IR From Visit 1 to Visit 2
Description: Investigators will measure the change in glycemic measures between Visit 1 (Day 1) and Visit 2 (Day 8) as an index of Metformin response, and compare them by genotype at selected loci. HOMA-IR is calculated from fasting glucose and fasting insulin values at both visit 1 (day 1) and visit 2 (day 8). HOMA-IR was calculated using (fasting glucose*fasting insulin)/405) formula. A bigger difference/drop between visit 1 and visit 2 will show that metformin had an effect on insulin resistance index for these participants. The higher the HOMA-IR, the more insulin resistant you are.
Time Frame: Day 1 (Visit 1) and Day 8 (Visit 2)
Population: We looked at HOMA-IR at Visit 2 minus HOMA-IR at visit 1 to see if there are differences by genotype at rs7903146 after Metformin treatment in the 1000 subjects in this study. 10 subjects didn't pass the QC for genotype analysis.
Measure: Mean (Standard Deviation); unit: (mg/dl*uU/ml²)
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 990
(mg/dl*uU/ml²)
  HOMA-IR Visit 1 - HOMA IR Visit 2 in CC Gentoype: number analyzed (Participants) | 500
  HOMA-IR Visit 1 - HOMA IR Visit 2 in CC Gentoype | 0.09 (1.9)
  HOMA-IR Visit 1 - HOMA IR Visit 2 in CT Gentoype: number analyzed (Participants) | 400
  HOMA-IR Visit 1 - HOMA IR Visit 2 in CT Gentoype | 0.04 (1.98)
  HOMA-IR Visit 1 - HOMA IR Visit 2 in TT Gentoype: number analyzed (Participants) | 90
  HOMA-IR Visit 1 - HOMA IR Visit 2 in TT Gentoype | -0.45 (0.29)

5. Secondary Outcome: Incretin Levels
Description: Investigators will measure GLP-1 and GIP during the OGTT from 0 to 120 minutes of Visit 2, and compare them by genotype at selected loci.
Time Frame: 0, 5, 10, 15, 30, 60 and 120 minutes, Day 8 (Visit 2)
Population: We only measured GLP-1 and GIP in a subset of the study population. We are showing Area under the curve results for GLP-1 total, GLP-1 active, and GIP by genotype at rs7903146 in TCF7L2.
Measure: Mean (Standard Deviation); unit: pmol/L x time (minutes)
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 168
pmol/L x time (minutes)
  GLP-1 Total AUC at CC genotype: number analyzed (Participants) | 60
  GLP-1 Total AUC at CC genotype | 1176.2 (523)
  GLP-1 Total AUC at CT genotype: number analyzed (Participants) | 56
  GLP-1 Total AUC at CT genotype | 1286.4 (540.4)
  GLP-1 Total AUC at TT genotype: number analyzed (Participants) | 52
  GLP-1 Total AUC at TT genotype | 1749.3 (1399)
  GLP-1 Active AUC at CC genotype: number analyzed (Participants) | 60
  GLP-1 Active AUC at CC genotype | 879 (316.6)
  GLP-1 Active AUC at CT genotype: number analyzed (Participants) | 56
  GLP-1 Active AUC at CT genotype | 1060.8 (687.3)
  GLP-1 Active AUC at TT genotype: number analyzed (Participants) | 52
  GLP-1 Active AUC at TT genotype | 1415.7 (1681.2)
  GIP AUC at CC genotype: number analyzed (Participants) | 60
  GIP AUC at CC genotype | 23523 (8227)
  GIP AUC at CT genotype: number analyzed (Participants) | 56
  GIP AUC at CT genotype | 24041.2 (8126)
  GIP AUC at TT genotype: number analyzed (Participants) | 52
  GIP AUC at TT genotype | 20183.1 (5892.8)

6. Secondary Outcome: Proinsulin (Fasting) at Visit 1 and Visit 2 by Genotype for rs7903146
Description: Investigators will measure proinsulin levels at regular intervals during Visits 1 and 2, and compare them by genotype at selected loci.
Time Frame: Day 1 (Visit 1) and Day 8 (Visit 2)
Population: Fasting Proinsulin were measured only in a subset of study samples. We are showing fasting data at Day 1, Visit 1 and Day 8, Visit 2 by genotype at rs7903146 (in TCF7L2).
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 589
pmol/L
  ProInsulin at Visit 1 at CC Genotype: number analyzed (Participants) | 300
  ProInsulin at Visit 1 at CC Genotype | 20.5 (21.2)
  ProInsulin at Visit 1 at CT Genotype: number analyzed (Participants) | 238
  ProInsulin at Visit 1 at CT Genotype | 23.4 (25.2)
  ProInsulin at Visit 1 at TT Genotype: number analyzed (Participants) | 51
  ProInsulin at Visit 1 at TT Genotype | 25.1 (21.2)
  ProInsulin at Visit 2 at CC Genotype: number analyzed (Participants) | 300
  ProInsulin at Visit 2 at CC Genotype | 19.4 (21.6)
  ProInsulin at Visit 2 at CT Genotype: number analyzed (Participants) | 238
  ProInsulin at Visit 2 at CT Genotype | 19.1 (19)
  ProInsulin at Visit 2 at TT Genotype: number analyzed (Participants) | 51
  ProInsulin at Visit 2 at TT Genotype | 21.4 (20.9)

7. Secondary Outcome: Metabolomics
Description: Investigators will perform metabolomic profiling of plasma samples at regular intervals during Visits 1 and 2, by using initially a targeted approach on an existing platform that measures ~400 metabolites (both polar and non-polar); they will compare their relative concentrations by genotype at selected loci before and after the study interventions.
Time Frame: Day 1 (Visit 1) and Day 8 (Visit 2)
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Vitamin D
Description: Investigators will measure 25-hydroxy vitamin D levels at baseline, and examine its effects on glycemic measures during Visits 1 and 2.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Fasting Glucagon at Visit 1 and Visit 2 by Genotype for rs7903146
Description: Investigators will measure glucagon levels at regular intervals during Visits 1 and 2, and compare them by genotype at selected loci.
Time Frame: Day 1 (Visit 1) and Day 8 (Visit 2)
Population: Fasting glucagon were measured only in a subset of study samples. We are showing fasting data at Day 1, Visit 1 and Day 8, Visit 2 by genotype at rs7903146 (in TCF7L2).
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Glipizide and Metformin
Number analyzed (Participants) | 556
pg/ml
  Glucagon at Visit 1 at CC Genotype: number analyzed (Participants) | 286
  Glucagon at Visit 1 at CC Genotype | 29.9 (18.0)
  Glucagon at Visit 1 at CT Genotype: number analyzed (Participants) | 226
  Glucagon at Visit 1 at CT Genotype | 28.4 (19.7)
  Glucagon at Visit 1 at TT Genotype: number analyzed (Participants) | 44
  Glucagon at Visit 1 at TT Genotype | 25.7 (16.3)
  Glucagon at Visit 2 at CC Genotype: number analyzed (Participants) | 286
  Glucagon at Visit 2 at CC Genotype | 28.4 (16.4)
  Glucagon at Visit 2 at CT Genotype: number analyzed (Participants) | 226
  Glucagon at Visit 2 at CT Genotype | 28 (15.9)
  Glucagon at Visit 2 at TT Genotype: number analyzed (Participants) | 44
  Glucagon at Visit 2 at TT Genotype | 28.5 (17.5)

ADVERSE EVENTS:
Time Frame: 8 days (on day 1 the subjects had their first study visit and their second study visit was on day 8).
Arm/Group | Glipizide and Metformin
All-Cause Mortality (participants affected / at risk) | 0/1033
Serious Adverse Events (participants affected / at risk) | 0/1033
Other Adverse Events (participants affected / at risk) | 0/1033

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes